CLINICAL TRIAL: NCT02740413
Title: TREATMENT PATTERNS AND OUTCOMES IN PATIENTS TREATED WITH BENEFIX OR REFACTO/REFACTO AF - A SWEDISH COHORT STUDY
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1821054; NCT02740413 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2015-12-16; First posted 2016-04-15 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Haemophilia A: Patients in The MHR diagnosed with Haemophilia A
- Patients with Haemophilia B: Patients in The MHR diagnosed with Haemophilia B

SUMMARY:
The overall aim of the study is to describe demographic and clinical characteristics, treatment patterns and outcomes, in the populations of hemophilia patients treated with BeneFIX and ReFacto/ReFacto AF in Sweden

DETAILED DESCRIPTION:
The overall aim of the study is to describe demographic and clinical characteristics, treatment patterns and outcomes, as well as the related direct treatment costs in the populations of hemophilia patients treated with BeneFIX and ReFacto/ReFacto AF, and in subgroups (e.g. level of severity) at the MHC in Sweden.

The study population will consist of all patients diagnosed with haemophilia (D66.9 (haemophilia A) D67.9 (haemophilia B) in International Statistical Classification of Diseases and Related Health Problems (ICD-10) that have been registered in the MHR since 1977 and that have had at least one registered prescription of BeneFIX or ReFacto/ReFacto AF in the MHR since market authorization of the respective product (Benefix August 27 1997, ReFacto April 13 1999, ReFacto AF July 1 2009). Diseased individuals are included. Information on drugs picked up at the pharmacy is available in the Prescribed Drug Register from 2005.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of all patients diagnosed with hemophilia (D66.9 (hemophilia A) D67.9 (hemophilia B) in International Statistical Classification of Diseases and Related Health Problems (ICD-10) that have been registered in the Malmö Hemophilia Register since 1977 and that have had at least one registered prescription of BeneFIX or ReFacto/ReFacto AF in the MHR since market authorization of the respective product

Exclusion Criteria:

* No exclusion criteria in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of all patients diagnosed with hemophilia (D66.9 (hemophilia A) D67.9 (hemophilia B) in International Statistical Classification of Diseases and Related Health Problems (ICD-10) that have been registered in the Malmö Hemophilia Register since 1977 and that have had at least one registered prescription of BeneFIX or ReFacto/ReFacto AF in the MHR since market authorization of the respective product (Benefix August 27 1997, ReFacto April 13 1999, ReFacto AF July 1 2009). Diseased individuals are included.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1821054

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was a retrospective population-based register study. Detailed data on each participant diagnosed with haemophilia was retrieved from the Malmö Haemophilia Register (MHR) in January 2016 covering the period of January 2005 up to December 2015.
Groups:
- Benefix/Refacto/Refacto AF: Participants diagnosed with haemophilia A and B who were registered in the MHR and had at least one registered prescription of Benefix or Refacto/Refacto AF were included in the study and their data (for the duration of 11 years, i.e. 2005-2015) was retrospectively observed.
Period: Overall Study
Arm/Group | Benefix/Refacto/Refacto AF
Started | 86
Completed | 86
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: MHR Benefix or Refacto/Refacto AF analysis set: all participants diagnosed with haemophilia A or B in International Statistical Classification of Diseases and Related Health Problems (ICD-10), registered in MHR since 1977, had at least 1 registered prescription of Benefix or Refacto/Refacto AF in MHR since market authorization of respective product
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (20.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Year of Birth for Participants [Median (Full Range); unit: years] | 1985 [1932 to 2012]
Percentage of Participants Who Had Died During the Prior 11 Year Period [Number; unit: percentage of participants] | 0
Percentage of Participants With Severe, Moderate and Mild Haemophilia A or B [Number; unit: percentage of participants] — Criteria for severity was defined as MHR standard categories Mild: factor (VIII and IX) level 5-40 percent (%); Moderate: factor level 1-5% and Severe: factor level less than 1%.
  percentage of participants
    Mild | 20
    Moderate | 24
    Severe | 56
Percentage of Participants with Inhibitor Status [Number; unit: percentage of participants] — Participants who developed inhibitory antibodies against factor VIII or IX were analyzed and their inhibitor status were categorized as: current, ever or never, based on last available observation in the MHR. Criteria for inhibitor development was as: if noted yes in the MHR at the date of data extraction: current; if noted yes at an earlier date: ever; if never noted yes in the MHR: never.
  percentage of participants
    Current | 2
    Ever | 1
    Never | 97
Percentage of Participants Infected With Hepatitis C [Number; unit: percentage of participants] — Participants categorized as Hepatitis-C positive based on last available observation in the MHR.
  percentage of participants | 40
Percentage of Participants With Positive Human Immunodeficiency Virus (HIV) status [Number; unit: percentage of participants] — Participants categorized as HIV positive based on last available observation in the MHR.
  percentage of participants | 5

OUTCOME MEASURES:

1. Primary Outcome: Age of Participants at Disease Diagnosis
Time Frame: At disease diagnosis within 11 years before the study start date (Day 1)
Population: MHR Benefix or Refacto/Refacto AF analysis set: all participants diagnosed with haemophilia A or B in ICD-10, registered in MHR since 1977, had at least 1 registered prescription of Benefix or Refacto/Refacto AF in MHR since market authorization of respective product. Here, "N"= number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: years
Groups:
- Benefix/Refacto/Refacto AF: Haemophilia A: Participants diagnosed with haemophilia A who were registered in the MHR and had at least one registered prescription of Benefix or Refacto/Refacto AF were included in the study and their data (for the duration of 11 years, i.e. 2005-2015) was retrospectively observed.
- Benefix/Refacto/Refacto AF: Haemophilia B: Participants diagnosed with haemophilia B who were registered in the MHR and had at least one registered prescription of Benefix or Refacto/Refacto AF were included in the study and their data (for the duration of 11 years, i.e. 2005-2015) was retrospectively observed.
Arm/Group | Benefix/Refacto/Refacto AF: Haemophilia A | Benefix/Refacto/Refacto AF: Haemophilia B
Number analyzed (Participants) | 28 | 50
years | 5 (10.1) | 7 (10.7)

2. Primary Outcome: Age of Participants at Start of Treatment With Benefix or Refacto
Time Frame: At start of treatment with Benefix/Refacto within 11 years before the study start date (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Benefix/Refacto/Refacto AF: Haemophilia A | Benefix/Refacto/Refacto AF: Haemophilia B
Number analyzed (Participants) | 32 | 52
years | 18 (16.2) | 30 (20.9)

3. Primary Outcome: Age of Participants at Start of Replacement Treatment
Description: Participants diagnosed with coagulation disorders received intravenous replacement treatment of the missing coagulation factor. Replacement treatment could be given prophylactically or to stop the bleed and/or to stop it from becoming more severe.
Time Frame: At start of replacement treatment within 11 years before the study start date (Day 1)
Population: MHR Benefix or Refacto/Refacto AF analysis set: all participants diagnosed with haemophilia A or B in ICD-10, registered in MHR since 1977, had at least 1 registered prescription of Benefix or Refacto/Refacto AF in MHR since market authorization of respective product.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Benefix/Refacto/Refacto AF: Haemophilia A | Benefix/Refacto/Refacto AF: Haemophilia B
Number analyzed (Participants) | 33 | 53
years | 16 (15.6) | 27 (20.3)

4. Primary Outcome: Average Prescribed Dose Per Infusion for Factor VIII and Factor IX Concentrates
Description: Participants diagnosed with coagulation disorders received intravenous replacement treatment of the missing coagulation factor (Factor VIII or IX). Data was measured in international units (IU) for factor VIII and factor IX concentrates.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: MHR Benefix or Refacto/Refacto AF analysis set: all participants diagnosed with haemophilia A or B in ICD-10, registered in MHR since 1977, had at least 1 registered prescription of Benefix or Refacto/Refacto AF in MHR since market authorization of respective product. Here, "n"= number of participants with available data for each category.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
IU
  Factor VIII: number analyzed (Participants) | 31
  Factor VIII | 1600 (700)
  Factor IX: number analyzed (Participants) | 50
  Factor IX | 2500 (900)

5. Primary Outcome: Average Prescribed Dose Per Kilogram Bodyweight for Factor VIII and Factor IX Concentrates
Description: The average dose per kilogram body weight of factor VIII and IX was defined as a set of two derived variables from the MHR based on information on prescribed replacement treatment (Benefix or Refacto/Refacto AF): prescribed dose per infusion divided by registered body weight (all participants) and prescribed dose per week (prescribed dose per infusion multiplied by registered number of infusions per week) divided by registered body weight (only participants on prophylaxis).
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: IU per kilogram
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
IU per kilogram
  Factor VIII: number analyzed (Participants) | 29
  Factor VIII | 27 (10)
  Factor IX: number analyzed (Participants) | 50
  Factor IX | 37 (11)

6. Primary Outcome: Percentage of Participants on Prophylactic Treatment
Description: Prophylactic treatment was defined as administration of drug regularly to reduce the insufficiency of coagulation factor to prevent bleeding to occur.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Benefix/Refacto/Refacto AF: Haemophilia A | Benefix/Refacto/Refacto AF: Haemophilia B
Number analyzed (Participants) | 33 | 53
percentage of participants | 78 | 56

7. Primary Outcome: Average Prescribed Frequency of Infusions Per Week Dispensed for Haemophilia A or B Participants With Prophylaxis
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: MHR Benefix or Refacto/Refacto AF analysis set: all participants diagnosed with haemophilia A or B in ICD-10, registered in MHR since 1977, had at least 1 registered prescription of Benefix or Refacto/Refacto AF in MHR since market authorization of respective product. Here, "N"= number of participants with prophylaxis.
Measure: Mean (Standard Deviation); unit: infusions per week
Arm/Group | Benefix/Refacto/Refacto AF: Haemophilia A | Benefix/Refacto/Refacto AF: Haemophilia B
Number analyzed (Participants) | 25 | 28
infusions per week | 3.9 (1.6) | 3.1 (2.4)

8. Primary Outcome: Average Prescribed Annual Dose of Factor VIII and IX Concentrates for Participants on Prophylaxis
Description: Participants diagnosed with coagulation disorders received intravenous replacement treatment of the missing coagulation factor (Factor VIII or IX). Prescribed annual dose of factor concentrate was derived from the MHR registration of prescribed annual dose of factor concentrate.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: Analysis was performed on MHR Benefix or Refacto/Refacto AF analysis set. Here, "overall number of participants analysed" signifies participants who were evaluable for this outcome measure and "number analysed" signifies number of participants with available data for each category.
Measure: Mean (Standard Deviation); unit: IU/year
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 53
IU/year
  Factor VIII: number analyzed (Participants) | 21
  Factor VIII | 286000 (116000)
  Factor IX: number analyzed (Participants) | 20
  Factor IX | 367000 (187000)

9. Primary Outcome: Average Prescribed Annual Dose of Factor VIII and IX Concentrates Per Kilogram Bodyweight for Participants on Prophylaxis
Description: Participants diagnosed with coagulation disorders received intravenous replacement treatment of the missing coagulation factor (Factor VIII or IX). Prescribed annual dose of factor concentrate per kilogram body weight was derived from the MHR registration of prescribed annual dose of factor concentrate and the registered body weight.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: IU/kg/year
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 53
IU/kg/year
  Factor VIII: number analyzed (Participants) | 20
  Factor VIII | 4500 (800)
  Factor IX: number analyzed (Participants) | 20
  Factor IX | 4700 (2200)

10. Primary Outcome: Average Annual Registered Consumption of Factor VIII and IX Concentrates
Description: Participants diagnosed with coagulation disorders received intravenous replacement treatment of the missing coagulation factor (Factor VIII or IX). Average annual registered consumption of factor VIII and IX concentrates was defined as MHR registered participant's reports on factor concentrate consumption during calendar year.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/year
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 8
IU/year
  Factor VIII | 80000 (70000)
  Factor IX | 73000 (53000)

11. Primary Outcome: Number of Participants With Consumption of Factor VIII, Factor IX, Factor rVIIa and/or aPCC Concentrate
Description: Participants who develop inhibitors to factor VIII or IX concentrates were treated with bypassing agents in the form of activated prothrombin complex concentrate (aPCC) which was measured in units (U) and/or recombinant factor VIIa (rFVIIa) measured in micrograms (mcg).
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
Participants
  Factor VIII | 33
  Factor IX | 53
  Factor rVIIa | 0
  Factor aPCC | 0

12. Primary Outcome: Percentage of Time on Refacto or Benefix
Description: Percentage of time (in days) on Refacto/Refacto AF or Benefix was calculated as total number of days when participant was prescribed Refacto/Refacto AF or Benefix over the total number of days on any replacement treatment. Total number of days on any replacement treatment was derived from date of start of replacement treatment according to MHR and August 31, 2015 or date of death, whichever was earliest.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 76
days
  Percentage of time on Refacto | 0 [0 to 100]
  Percentage of time on Benefix | 19 [0 to 100]

13. Primary Outcome: Average Use of Factor Concentrate Per Surgery Event at Hospital for Invasive Procedures
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU per surgery event
Arm/Group | Benefix/Refacto/Refacto AF: Haemophilia A | Benefix/Refacto/Refacto AF: Haemophilia B
Number analyzed (Participants) | 33 | 53
IU per surgery event | 13447 (10695) | 24171 (20976)

14. Primary Outcome: Average Factor Concentrate Use at Hospital for Invasive Procedures
Description: Average factor concentrate use was calculated as percentage of total annual use of factor concentrates (in IU) at hospital for invasive procedures.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of factor concentrate
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
percentage of factor concentrate | 2 (14)

15. Primary Outcome: Average Annual Number of Filled Prescriptions of Factor Concentrate
Description: Data at end of every year was based on the number of filled prescriptions during the last 3 years.
Time Frame: For a duration of 3 years (for up to 11 years before the study start Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: prescriptions
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
prescriptions
  2005: number analyzed (Participants) | 50
  2005 | 5 (4)
  2008: number analyzed (Participants) | 53
  2008 | 11 (8)
  2011: number analyzed (Participants) | 63
  2011 | 11 (7)
  2014: number analyzed (Participants) | 62
  2014 | 11 (7)

16. Primary Outcome: Average Annual Number of Dispensed Units of Factor Concentrate
Description: To assess annual consumption of factor concentrates, calculations were based on prescription date as start of use and the day before the next prescription as the last date of use of the factor concentrates retrieved. The annual number of dispensed units of factor concentrate were then summed up of all dispensed units of factor concentrate with periods within the calendar year plus estimates of average daily use periods extending over two years. Data at end of every year was based on the number of dispensed units of factor concentrate during the last 3 years.
Time Frame: For a duration of 3 years (for up to 11 years before the study start Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: dispensed units
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
dispensed units
  Factor VIII (2005): number analyzed (Participants) | 22
  Factor VIII (2005) | 109000 (79000)
  Factor VIII (2008): number analyzed (Participants) | 23
  Factor VIII (2008) | 219000 (151000)
  Factor VIII (2011): number analyzed (Participants) | 24
  Factor VIII (2011) | 220000 (138000)
  Factor VIII (2014): number analyzed (Participants) | 25
  Factor VIII (2014) | 235000 (130000)
  Factor IX (2005): number analyzed (Participants) | 26
  Factor IX (2005) | 68000 (71000)
  Factor IX (2008): number analyzed (Participants) | 28
  Factor IX (2008) | 163000 (140000)
  Factor IX (2011): number analyzed (Participants) | 36
  Factor IX (2011) | 194000 (217000)
  Factor IX (2014): number analyzed (Participants) | 34
  Factor IX (2014) | 212000 (200000)

17. Primary Outcome: Average Number of Units of Benefix or Refacto
Description: Data from the National Board of Health and Welfare (NBHW) had information on all filled prescriptions from July 1, 2005-last date of observation (August 31, 2015). Derived variable calculated as total number of units of filled prescriptions of Refacto/Refacto AF and Benefix over the total units of all factor VIII concentrates and factor IX concentrates, respectively. Total number of units were derived from the date of start of NBHW to last available observation or date of death, whichever was earliest.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
units
  Refacto - Factor VIII: number analyzed (Participants) | 22
  Refacto - Factor VIII | 229000 (130000)
  Benefix - Factor IX: number analyzed (Participants) | 28
  Benefix - Factor IX | 191000 (163000)

18. Primary Outcome: Total Number of Bleeds
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bleeds
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 33
bleeds | 1.1 (1.4)

19. Primary Outcome: Number of Joint Bleed, Muscle Bleeds and Other Bleed Events in Participants
Description: Joint bleeds included traumatic and spontaneous joint bleeds, muscle bleeds included traumatic and spontaneous soft tissue bleeds and other bleed events included intracranial bleed, gastrointestinal bleed and urinary tract bleed.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 3
Measure: Number; unit: bleeds
Units Other Than Participants: bleeds
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
Number analyzed (bleeds) | 279
bleeds
  Joint bleed | 68
  Muscle bleed | 179
  Other bleed | 32

20. Primary Outcome: Gilbert Joint Score
Description: Gilbert joint score was an instrument to measure joint health in the domain of body structure and function (i.e. impairment), of the joints most commonly affected by bleeding in haemophilia - knees, ankles, elbows. Total score ranged from 0-100, evaluating ankle, knee and elbow, where "0" indicated normal joint function, "100" indicated worst joint function, where higher values indicated more impairment in joints.
Time Frame: Data analyzed on study start Day 1 for the duration of 4 years (2005 to 2009)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 59
scores on a scale | 6 (8)

21. Primary Outcome: Haemophilia Joint Health Score
Description: Haemophilia Joint Health Score (HJHS) was used to assess joint damage in participants with haemophilia. Total score ranges from 0 to 124, where, 0 indicates normal function, and 124 indicates worst joint function, higher values indicated more damage in joints.
Time Frame: Data analyzed on study start Day 1 for the duration of 6 years (2009 to 2015)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 75
scores on a scale | 15 (17)

22. Primary Outcome: Percentage of Participants With Surgeries
Description: Percentage of participants who had any type of surgery (arthrodesis, surgery on foot, nose, elbow, hand or shoulder, surgery on hip, surgery on knee, tooth extraction, venous port or any other) during the data observation period were reported.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
percentage of participants
  Arthrodesis | 8
  Surgery on foot, nose, elbow, hand or shoulder | 8
  Surgery on hip | 7
  Surgery on knee | 11
  Tooth extraction | 17
  Venous port | 15
  Other surgeries | 34

23. Primary Outcome: Average Relative Dose Intensity of Factor Concentrate Dispensed for Haemophilia A or B Participants on Prophylaxis Based on Dispensed Volume of Units
Description: Relative dose intensity based on dispensed volume of units was calculated using annual dispensed volume of factor concentrate per participant divided by annual prescribed dose per participant. Data was analysed for 2 categories separately: children/adolescents and adults.
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of factor concentrate
Groups:
- Haemophilia A: Participants with haemophilia A registered in the Malmo Haemophilia Register (MHR) with at least one prescription of BeneFIX and ReFacto/ReFacto AF were observed for 11 years (2005-2015).
- Haemophilia B: Participants with haemophilia B registered in the Malmo Haemophilia Register (MHR) with at least one prescription of BeneFIX and ReFacto/ReFacto AF were observed for 11 years (2005-2015).
Arm/Group | Haemophilia A | Haemophilia B
Number analyzed (Participants) | 33 | 53
percentage of factor concentrate
  Children/Adolescents: number analyzed (Participants) | 11 | 13
  Children/Adolescents | 103 (33) | 96 (22)
  Adults: number analyzed (Participants) | 22 | 40
  Adults | 88 (24) | 71 (33)

24. Secondary Outcome: Average Annual Cost of Prescribed Factor Concentrate and Dispensed Replacement Treatment
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: SEK
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
SEK
  Prescribed Factor Concentrate: number analyzed (Participants) | 39
  Prescribed Factor Concentrate | 2085000 (875000)
  Dispensed Replacement Treatment: number analyzed (Participants) | 59
  Dispensed Replacement Treatment | 1351000 (944000)

25. Primary Outcome: Average Cost of Replacement Treatment (Benefix or Refacto/Refacto AF) Related to Bleed Event
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Swedish Krona (SEK)
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 13
Swedish Krona (SEK) | 100000 (121000)

26. Secondary Outcome: Average Cost of Replacement Treatment Related to Invasive Procedures
Time Frame: For the duration of 11 years before the study start date (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SEK
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 9
SEK | 71000 (72000)

27. Other Pre Specified Outcome: Average Annual Cost of Replacement Treatment Related to Invasive Procedures
Time Frame: Data analyzed on study start Day 1 for Year 1 (2005) and Year 7 (2011)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: SEK
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
SEK
  2005: number analyzed (Participants) | 9
  2005 | 165000 (143000)
  2011: number analyzed (Participants) | 5
  2011 | 63000 (51000)

28. Other Pre Specified Outcome: Average Cost for Replacement Treatment Related to Invasive Procedures
Description: The average cost for replacement treatment related to invasive procedures was derived from the percentage of total costs for dispensed replacement therapy and calculated as: cost of factor concentrate used for invasive procedures/ total cost of factor concentrate.
Time Frame: Data analyzed on study start Day 1 for Year 1 (2005) and Year 7 (2011)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of cost
Arm/Group | Benefix/Refacto/Refacto AF
Number analyzed (Participants) | 86
percentage of cost
  2005: number analyzed (Participants) | 8
  2005 | 124 (245)
  2011: number analyzed (Participants) | 5
  2011 | 14 (21)

ADVERSE EVENTS:
Time Frame: Within 11 years (from 2005 to 2015) before the study start date (Day 1)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Benefix/Refacto/Refacto AF
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-06-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT02740413/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT02740413/SAP_001.pdf